CLINICAL TRIAL: NCT02509780
Title: The Mineral Water of Vichy and the Urinary Alkalization: A Study of the Dose - Effect of Bicarbonate Salt Water on the Urinary pH in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Jean-Marie De Meyer, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUB-Vichy
Record Dates: First submitted 2015-07-22; First posted 2015-07-28 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Vichy; urine alkalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vichy (Experimental)
  Interventions: Other: Vichy

INTERVENTIONS:
Other: Vichy — Volunteers will be asked during 3 days to take their usual intake of fluids. For the following 7 days, they will take the usual intake of fluids plus 250 ml of Vichy water at 1 pm. For the following 7 days, they will take the usual intake of fluids plus 250 ml of Vichy water at 7 am and 7 pm. Ph and density measurement of urine will be made three times a day, at 7 am, 2 pm and 8 pm.

SUMMARY:
Vichy water is a type of spring water which traditionally comes from the famous spa town of Vichy, France. The springs which feed Vichy carry a high amount of dissolved minerals. Alkaline salts such as sodium bicarbonate are a primary ingredient in Vichy water, along with calcium and magnesium carbonates.

Bicarbonates alkalinize urine, which is fundamental in preventing and/or diluting uric acid crystals. These are the main component of the uric acid stones or even oxalate stones, which generally " use " a crystal of uric acid as nucleus for stone formation. Cystine stones can also be treated by alkalinizing urine.

Any disorder leading to a low urinary pH ( < 5.5 ) may predispose to stone formation. In this context , the solution of uric acid and the prevention and treatment of uric acid stones can be obtained by alkalization of the urine . The ideal alkalization is achieved when a urinary pH of 6-6.5 can be reached.

The aim of this study is to evaluate the quantity of daily intake of the Vichy water necessary to obtain this alkalization of the urine. There are no data available in the literature about the relationship between the absolute quantity of Vichy water taken and the urinary pH ; nor about the possible influence of the Body Mass Index on this relationship.

DETAILED DESCRIPTION:
Vichy water is a type of spring water which traditionally comes from the famous spa town of Vichy, France. The springs which feed Vichy carry a high amount of dissolved minerals, and they create a distinctive naturally effervescent bubbling water. Alkaline salts such as sodium bicarbonate are a primary ingredient in Vichy water, along with calcium and magnesium carbonates. The water is sometimes slightly odorous, with substances like sulfur naturally bubbling up with the water. The water also has a distinct taste, due to the dissolved minerals.

Bicarbonates alkalinize urine, which is fundamental in preventing and/or diluting uric acid crystals. These are the main component of the uric acid stones or even oxalate stones , which generally " use " a crystal of uric acid as nucleus for stone formation. Cystine stones can also be treated by alkalinizing urine.

Three conditions influence the potential for uric acid stone formation : the quantitative excretion of uric acid , the volume of urine as it affects the urinary concentration of uric acid, and the urinary pH which seems to be the most important pathogenic factor . Uric acid is a weak acid with a pKa of 5.35 at 37° C . At that pH , half of the uric acid is present as the urate salt and half as free uric acid . Because sodium urate is approximately 20 times more soluble than the free acid, the relative proportion present as free uric acid strongly determinates the risk of stone formation . Low urinary pH increases concentrations of sparingly soluble undissociated uric acid, which leads to direct precipitation of uric acid .

Any disorder leading to a low urinary pH ( < 5.5 ) may predispose to stone formation. For example a chronic metabolic acidosis can lead to a low urinary pH, a hypercalciuria and a hypocitraturia . "Gouty diathesis " refers to a stone - forming propensity characterized by low urinary pH of unknown etiology with or without associated gouty arthritis.

In this context , the solution of uric acid and the prevention and treatment of uric acid stones can be obtained by alkalization of the urine. The ideal alkalization is achieved when a urinary pH of 6-6.5 can be reached.

The aim of this study is to evaluate the quantity of daily intake of the Vichy water necessary to obtain this alkalization of the urine. There are no data available in the literature about the relationship between the absolute quantity of Vichy water taken and the urinary pH ; nor about the possible influence of the Body Mass Index on this relationship.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 50 years of age
* Available to participate for the planned duration of the study
* Able and willing to complete the study process

Exclusion Criteria:

* Renal disease
* Diabetes
* Hypertension
* Heart failure

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Daily mean urine pH value (normal intake of fluids) | Day 1
  The study starts with a 3 days "running" period with usual intake of fluids. Each study day three samples of urine are collected for pH measurement with a pH indicator stick ( at 7 am, at 2 pm , and at 8 pm ), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (250 ml Vichy) | Day 4
  After the three days running period, a 7 days period is observed with usual intake of fluids plus 250 ml of Vichy water at 1 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick ( at 7 am, at 2 pm and at 8 pm), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (500 ml Vichy) | Day 11
  Afterwards follows a 7 days period with usual intake of fluids plus 500 ml of Vichy water, divided in two doses: one intake at 7am and one intake at 7 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick (at 7 am, at 2 pm , and at 8 pm ), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (normal intake of fluids) | Day 2
  The study starts with a 3 days "running" period with usual intake of fluids. Each study day three samples of urine are collected for pH measurement with a pH indicator stick ( at 7 am, at 2 pm , and at 8 pm ), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (normal intake of fluids) | Day 3
  The study starts with a 3 days "running" period with usual intake of fluids. Each study day three samples of urine are collected for pH measurement with a pH indicator stick ( at 7 am, at 2 pm , and at 8 pm ), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (250 ml Vichy) | Day 5
  After the three days running period, a 7 days period is observed with usual intake of fluids plus 250 ml of Vichy water at 1 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick ( at 7 am, at 2 pm and at 8 pm), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (250 ml Vichy) | Day 6
  After the three days running period, a 7 days period is observed with usual intake of fluids plus 250 ml of Vichy water at 1 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick ( at 7 am, at 2 pm and at 8 pm), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (250 ml Vichy) | Day 7
  After the three days running period, a 7 days period is observed with usual intake of fluids plus 250 ml of Vichy water at 1 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick ( at 7 am, at 2 pm and at 8 pm), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (250 ml Vichy) | Day 8
  After the three days running period, a 7 days period is observed with usual intake of fluids plus 250 ml of Vichy water at 1 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick ( at 7 am, at 2 pm and at 8 pm), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (250 ml Vichy) | Day 9
  After the three days running period, a 7 days period is observed with usual intake of fluids plus 250 ml of Vichy water at 1 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick ( at 7 am, at 2 pm and at 8 pm), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (250 ml Vichy) | Day 10
  After the three days running period, a 7 days period is observed with usual intake of fluids plus 250 ml of Vichy water at 1 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick ( at 7 am, at 2 pm and at 8 pm), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (500 ml Vichy) | Day 12
  Afterwards follows a 7 days period with usual intake of fluids plus 500 ml of Vichy water, divided in two doses: one intake at 7am and one intake at 7 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick (at 7 am, at 2 pm , and at 8 pm ), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (500 ml Vichy) | Day 13
  Afterwards follows a 7 days period with usual intake of fluids plus 500 ml of Vichy water, divided in two doses: one intake at 7am and one intake at 7 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick (at 7 am, at 2 pm , and at 8 pm ), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (500 ml Vichy) | Day 14
  Afterwards follows a 7 days period with usual intake of fluids plus 500 ml of Vichy water, divided in two doses: one intake at 7am and one intake at 7 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick (at 7 am, at 2 pm , and at 8 pm ), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (500 ml Vichy) | Day 15
  Afterwards follows a 7 days period with usual intake of fluids plus 500 ml of Vichy water, divided in two doses: one intake at 7am and one intake at 7 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick (at 7 am, at 2 pm , and at 8 pm ), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (500 ml Vichy) | Day 16
  Afterwards follows a 7 days period with usual intake of fluids plus 500 ml of Vichy water, divided in two doses: one intake at 7am and one intake at 7 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick (at 7 am, at 2 pm , and at 8 pm ), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.
Daily mean urine pH value (500 ml Vichy) | Day 17
  Afterwards follows a 7 days period with usual intake of fluids plus 500 ml of Vichy water, divided in two doses: one intake at 7am and one intake at 7 pm. Each study day three samples of urine are collected for pH measurement with a pH indicator stick (at 7 am, at 2 pm , and at 8 pm ), and density measurement. Daily mean pH value will be computed. A urine specific density test (comparing the density of urine to the density of water) is a simple method to verify that total fluid intake doesn't vary substantially between the different study periods.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Demeyer, MD, Principal Investigator — CHU Brugmann; Panagiotis DROLAPAS, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium